CLINICAL TRIAL: NCT05913167
Title: Comparison of Erector Spina and Transversus Abdominus Plan Blocks
Brief Title: Comparison of Erector Spina Plan Block and Trnsversus Abdominis Plan Block in Laparoscopic Nephrectomy: Prospective Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zehra Ipek ARSLAN, Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: LAPNEF2023
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-12

CONDITIONS: Laparoscopic Nephrectomy
Keywords: laparoscopy; nephrectomy; erector spina plan block; transversus abdominis plan block; morphine consumption; analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: erector spina and transversus abdominis plane blocks
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know which block was administered outcome assessors will not know which block was administered
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector spina plan block (Active Comparator): Erector spina plan block will be administered to the patients in this group.
  Interventions: Procedure: laparoscopic nephrectomy
- Transversus abdominis plan block (Active Comparator): Transversus abdominis plan block will be administered to the patients in this group.
  Interventions: Procedure: laparoscopic nephrectomy

INTERVENTIONS:
Procedure: laparoscopic nephrectomy — laparoscopic nephrectomy

SUMMARY:
Nephrectomy pain was higher. erector spina plan block and transversus abdominis plan block had shown to be effective in abdominal surgeries. This study aimed to compare these two bloc analgesic efficacy in laparoscopic nephrectomy patients. The primary aim is postoperative morphine consumption.

DETAILED DESCRIPTION:
Patients ASA 18-65 who will undergo laparoscopic nephrectomy are included in this prospective randomized clinical trial. Patients will be divided into two groups; erector spina and transversus abdominis plane block. Anesthesia will. induced with propofol, fentanyl, and rocuronium will be administered for muscle relaxation. Bispectral index monitoring will be used for monitorisation of the depth of anesthesia. Remifentanil was used during the whole procedure. the amount of consumption will be recorded. Patient-controlled device will be used with morphine. The postoperative morphine consumption will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 age
* patients undergoing laparoscopic nephrectomy
* ASA 1-3

Exclusion Criteria:

* <18- >65 < age
* patients undergoing open nephrectomy
* ASA 4-5

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative morphine consumption | 24 hour postoperatively
  morphine patient controlled analgesia was applied to the patients

SECONDARY OUTCOMES:
Peroperative remifentanil consumptions | peroperatively
  continious remifentanil infusion was applied
postoperative analgesia numeric rating scales | postoperative 24 hours
  patients will give numbers to their pain first hour, 6th hour and 24 th hour after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No